CLINICAL TRIAL: NCT04498208
Title: Immune System Modulation by Enhanced vs Standard Prehabilitation Program in Patients Undergoing Elective Major Surgery - a Prospective Monocentric Randomized Single-blinded Controlled Trial
Brief Title: Immune Modulation by Enhanced vs Standard Prehabilitation Program Before Major Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Brice Gaudilliere, Principal Investigator, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: IRB-57570
Record Dates: First submitted 2020-07-28; First posted 2020-08-04 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Surgery; Immune System and Related Disorders; Preoperative Care; Gastrointestinal Disease; Urological Disease; Gynecologic Disease; Thoracic Diseases
Keywords: Personalized program; Physical Activity; Stress-reduction; Cognition; Nutrition; inflammatory; immune response
MeSH Terms: conditions — Gastrointestinal Diseases; Urologic Diseases; Genital Diseases, Female; Thoracic Diseases; Motor Activity

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Personalized prehabilitation (Experimental): Patients will participate in a personalized health optimization program combining one-on-one coaching, tailored to each patient's physical, nutritional, well-being and cognitive status baseline. Prehabilitation will last from a minimum of 14 days to a maximum of 42 days before surgery
  Interventions: Behavioral: Physical Prehabilitation; Behavioral: Stress Reduction Prehabilitation; Behavioral: Cognitive Prehabilitation; Behavioral: Nutrition Prehabilitation
- Standard prehabilitation (No Intervention): Patients in the control group will be provided with standard instructions in a hard-copy form specific to prehabilitation before surgery associating physical, nutritional, stress-reduction and cognitive recommendations without any personalized coaching for at least 14 days prior to surgery.

INTERVENTIONS:
Behavioral: Physical Prehabilitation — First, an evaluation of patient's aerobic capacity, functional mobility, functional strength, ambulation, fall risk, and overall mobility will be done by a trained member of the research team. Based on their functional level and preexisting conditions, therapeutic exercises will be recommended to optimize their strength, endurance, flexibility, and functional mobility in preparation for surgery. Decisions about the interventions are based on the assessment, individual patient characteristics, environmental factors, surgical type, and monitoring of the client's response and progress. Weekly sessions are 30-45 minutes long to monitor the client's response and progress their program. Based on their response to exercise (evaluated also by 2 apps: Timed Walk App and Smart Metronome & Tuner App), re-evaluation via the assessments described above, change their plan of care (alter frequency, resistance, exercises) or discontinuation of treatment could be decided.
  Arms: Personalized prehabilitation
Behavioral: Stress Reduction Prehabilitation — Participants will have the opportunity to learn techniques for mindfulness that have been established to reduce stress and assist with pain management with a member of the research team. Patients will be offered to listen to audio recording of relaxation sessions. Each session contains a relaxation technique that the patient practices while listening to the recording. Then the technique is used the next as a baseline to introduce a new technique more advanced. For some patients who struggle with the techniques the program will be adapted. Patients will choose 2 or 3 techniques and work on them.
  Arms: Personalized prehabilitation
Behavioral: Cognitive Prehabilitation — Cognitive prehabilitation will consist on the daily use of Lumosity training program, an already existing free app built to increase memory skills. The program proposed by Lumosity is tailored to each patient. The use of Lumosity will be monitored at each in-person session. Patients will be expected to complete at least three 5-minute sessions of Lumosity training per day.
  Arms: Personalized prehabilitation
Behavioral: Nutrition Prehabilitation — Nutrition prehabilitation will involve transitioning the patient to the Mediterranean diet with targets regarding hydration and the proportion of fruits, vegetables, whole grains, and healthy fats the patient will consume in a given day. This nutritional program is flexible, and it allows for specific physician and nutritionist-recommended dietary needs to be incorporated. The patient is also given tools to encourage success in healthier eating, including recipes, sample menus, healthy restaurant options, meal kit options, and local CSA box options
  Arms: Personalized prehabilitation

SUMMARY:
Over 30 million surgeries are performed annually in the US. Up to 30% of surgical patients experience delayed surgical recovery, marked by prolonged post-surgical pain, opioid consumption, and functional impairment, which contributes $8 billion annually to US health care costs. Novel interventions that improve the resolution of pain, minimize opioid exposure, and accelerate functional recovery after surgery are urgently needed.

Multi-modal pre-operative optimization programs (or "prehab") integrating exercise, nutrition, and stress reduction have been shown to safely and effectively improve outcomes after surgery. However, no objective biological markers assess prehab effectiveness and are able to tailor prehab programs to individual patients. Surgery is a profound immunological perturbation, during which a complex network of innate and adaptive immune cells is mobilized to organize the recovery process of wound healing, tissue repair, and pain resolution. As such, the in-depth assessment of a patient's immune system before surgery is a promising approach to tailor prehab programs to modifiable biological markers associated with surgical recovery. The primary goal of this clinical trial is to determine the effect of a personalized prehab program on patients immunological status before surgery.

DETAILED DESCRIPTION:
The study design is a prospective monocenter single-blinded randomized controlled trial in patients undergoing elective major abdominal surgery.

* Patients will be recruited during the surgical consultation, at least 14 days prior to surgery. If they choose to enroll, they will undergo randomization on the day of enrollment.
* Prehabilitation (Day 0): personalized or standard prehabilitation program will be proposed to the patients for a period of 2 to 6 weeks. Immunological, nutritional, physical, cognitive, anxiety and quality of life status will be quantified at baseline by previously trained personnel.
* From the beginning (Day 0) to the end of the prehabilitation program (Day 14 to Day 42): every 7 days, a compliance questionnaire will be filled by phone, by a trained member of the research team blinded to the treatment arm of the study
* End of the prehabilitation period (Day 14 to Day 42): Immunological, nutritional, physical, cognitive and anxiety status after prehabilitation will be recorded by a trained member of the research team blinded to the treatment arm of the study.
* Surgery (Day S)
* Post operative period

  * From Day S (2 hours after surgery end) to discharge from the hospital, length of stay, pain and adverse clinical events will be measured and recorded.
  * Immunological status will be assessed at Day S+1 by blood draw.
  * Cognitive function, neuropathic pain and quality of life will be assessed at Day S + 30.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥ 18 years)
* Competent to provide informed consent
* Undergoing major elective surgery under general anesthesia in ≥14 days from enrollment (abdominal, thoracic, plastic and neurosurgeries).
* Fluent in English

Exclusion Criteria:

* Premorbid conditions or orthopedic impairments with contraindications to exercise
* Cognitive disabilities defined as evolutive neurological or neurodegenerative disease
* ASA score 4 or higher or patient under palliative care
* Illiteracy (inability to read the English language).
* Expected length of stay at hospital < 48 hours
* Patient under tutorship or curatorship
* Pregnant or breast-feeding woman
* Absence of informed consent or request to not participate to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2020-10-07 (Actual); Primary Completion 2024-04-21 (Actual); Study Completion 2024-04-21 (Actual)

PRIMARY OUTCOMES:
Composite immunological score | immediately preoperatively
  Composite immunological score containing a combination of blood immune cell frequencies and intracellular signaling responses. This score will be normalized to "baseline" (i.e. before prehabilitation) score for each patient.

SECONDARY OUTCOMES:
Proportion of compliant patients | immediately preoperatively
  Patient's compliance to prehabilitation programs will be evaluated using a modified Rehabilitation Adherence Measure scale, that will be filled by phone every 7 days during the prehabilitation program, i.e. 2 to 6 times by patient. Compliant patient will be defined by a mean score >= 8/10.
6 Min Walk Test | immediately preoperatively
  Changes in physical status will be examined using 6 Min Walk Test. The evaluation should be based on differences between pre- and post prehabilitation performance.
Timed Up and Go Test | immediately preoperatively
  Changes in physical status will be examined using Timed Up and Go Test. The evaluation should be based on differences between pre- and post prehabilitation performance.
Five Times Sit to Stand Test | immediately preoperatively
  Changes in physical status will be examined using Five Times Sit to Stand Test. The evaluation should be based on differences between pre- and post prehabilitation performance.
Wall Squat Test | immediately preoperatively
  Changes in physical status will be examined using Wall Squat Test. The evaluation should be based on differences between pre- and post prehabilitation performance.
Body Mass Index | immediately preoperatively
  Body Mass Index will be recorded. The evaluation should be based on differences between pre- and post prehabilitation performance
Amsterdam Preoperative Anxiety and Information Scale | immediately preoperatively
  Prevalence and global severity of anxiety will be evaluated using the APAIS (Amsterdam Preoperative Anxiety and Information Scale). The evaluation should be based on differences between pre- and post prehabilitation performance.
Pain Catastrophizing Scale | immediately preoperatively
  Prevalence and global severity of anxiety will be evaluated using the Pain Catastrophizing Scale. The evaluation should be based on differences between pre- and post prehabilitation performance.
Changes in diet | immediately preoperatively
  Mediterranean Diet Score will be collected. The evaluation should be based on differences between pre- and post prehabilitation performance. A high intake of Mediterranean foods: cereals, legumes, fruit, vegetables, fish, Mon-unsaturated fatty acids to Saturated fatty acids (M/S) ratio, and wine were scored positive (1) and a high intake of the non-Mediterranean foods: dairy and meat negative (0). The score ranged from 0 to 9 and the higher the score the better the compliance to a traditional Mediterranean diet.
Changes in cognitive functions | immediately preoperatively
  Cognitive functions will evaluated by the qMCI test. The evaluation should be based on differences between pre- and post prehabilitation performance.
Incidence of postoperative complications | Postoperatively through to 30 days after surgery
  Postoperative complications will be scored by the Comprehensive Complication Index. The Comprehensive Complication Index (CCI®) is based on the complication grading by Clavien-Dindo Classification and implements every occurred complication after an intervention. The overall morbidity is reflected on a scale from 0 (no complication) to 100 (death).
Postoperative pain | Postoperatively through to 7 days after surgery
  Pain scores will be assessed daily by the patient-reported Visual Analog Scale. Visual analog scale to assess the perceived stress on a horizontal, non-calibrated line of 10 cm, ranging from very low (0) to very high (10)
Cumulative opioid consumption | Postoperatively through to day 7
  Cumulative opioid consumption will be obtained from the patients' charts up to 7 days after surgery or discharge from hospital if earlier.
Neuropathic pain | 30 days after surgery
  Neuropathic pain will be measured by the Patient Reported Outcome Measurement Information System (PROMIS) Neuropathic Pain Quality scale (PROMIS-PQ-Neuro). The questionnaire contains 5 items questions. Scores are based on patient responses to questions about pain intensity. 0 indicates no pain; 5 indicates the most pain imaginable. The total score may be up to 25.
Hospital length of stay | 30 days after surgery
  Hospital length of stay assessed from patients' medical administrative data in days
Changes in quality of life | 30 days after surgery
  Quality of life evaluated thanks to the SF-36 scale is a 36-item patient-reported questionnaire that covers eight health domains: physical functioning (10 items), bodily pain (2 items), role limitations due to physical health problems (4 items), role limitations due to personal or emotional problems (4 items), emotional well-being (5 items), social functioning (2 items), energy/fatigue (4 items), and general health perceptions (5 items). Scores for each domain range from 0 to 100, with a higher score defining a more favorable health state. Results will be normalized on "baseline" (before prehab) scores.

CONTACTS AND LOCATIONS:
Overall Officials: Brice Gaudilliere, MD, PhD, Principal Investigator — Stanford University; Cindy Kin, MD, MS, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gaudilliere B, Fragiadakis GK, Bruggner RV, Nicolau M, Finck R, Tingle M, Silva J, Ganio EA, Yeh CG, Maloney WJ, Huddleston JI, Goodman SB, Davis MM, Bendall SC, Fantl WJ, Angst MS, Nolan GP. Clinical recovery from surgery correlates with single-cell immune signatures. Sci Transl Med. 2014 Sep 24;6(255):255ra131. doi: 10.1126/scitranslmed.3009701. PMID 25253674
- [Background] Aghaeepour N, Kin C, Ganio EA, Jensen KP, Gaudilliere DK, Tingle M, Tsai A, Lancero HL, Choisy B, McNeil LS, Okada R, Shelton AA, Nolan GP, Angst MS, Gaudilliere BL. Deep Immune Profiling of an Arginine-Enriched Nutritional Intervention in Patients Undergoing Surgery. J Immunol. 2017 Sep 15;199(6):2171-2180. doi: 10.4049/jimmunol.1700421. Epub 2017 Aug 9. PMID 28794234
- [Background] Fragiadakis GK, Gaudilliere B, Ganio EA, Aghaeepour N, Tingle M, Nolan GP, Angst MS. Patient-specific Immune States before Surgery Are Strong Correlates of Surgical Recovery. Anesthesiology. 2015 Dec;123(6):1241-55. doi: 10.1097/ALN.0000000000000887. PMID 26655308
- [Background] Barberan-Garcia A, Ubre M, Roca J, Lacy AM, Burgos F, Risco R, Momblan D, Balust J, Blanco I, Martinez-Palli G. Personalised Prehabilitation in High-risk Patients Undergoing Elective Major Abdominal Surgery: A Randomized Blinded Controlled Trial. Ann Surg. 2018 Jan;267(1):50-56. doi: 10.1097/SLA.0000000000002293. PMID 28489682
- [Background] Minnella EM, Awasthi R, Loiselle SE, Agnihotram RV, Ferri LE, Carli F. Effect of Exercise and Nutrition Prehabilitation on Functional Capacity in Esophagogastric Cancer Surgery: A Randomized Clinical Trial. JAMA Surg. 2018 Dec 1;153(12):1081-1089. doi: 10.1001/jamasurg.2018.1645. PMID 30193337
- [Derived] Cambriel A, Tsai A, Choisy B, Sabayev M, Hedou J, Shelton E, Singh K, Amar J, Badea V, Bruckman S, Ganio E, Einhaus J, Feyaerts D, Stelzer I, Sato M, Langeron O, Bonham TA, Gaudilliere D, Shelton A, Kin C, Gaudilliere B, Verdonk F. Immune Modulation by Personalized vs Standard Prehabilitation Before Major Surgery: A Randomized Clinical Trial. JAMA Surg. 2026 Jan 1;161(1):20-30. doi: 10.1001/jamasurg.2025.4917. PMID 41222945
- [Derived] Cambriel A, Tsai A, Choisy B, Sabayev M, Hedou J, Shelton E, Singh K, Amar J, Badea V, Bruckman S, Ganio E, Einhaus J, Feyaerts D, Stelzer I, Sato M, Langeron O, Bonham TA, Gaudilliere D, Shelton A, Kin C, Gaudilliere B, Verdonk F. Immune Modulation by Personalized vs. Standard Prehabilitation Before Major Surgery: A Randomized Controlled Trial. medRxiv [Preprint]. 2025 Jun 4:2025.06.03.25328894. doi: 10.1101/2025.06.03.25328894. PMID 40502574